CLINICAL TRIAL: NCT04933370
Title: Evaluating the Efficacy of Different Stimulation Paradigms in Neuromodulation
Brief Title: Neuromodulation Parameter Efficacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Health Services, Calgary (Other)
Responsible Party: Principal Investigator, Fady Girgis, Physician, Alberta Health Services, Calgary
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB21-0692
Record Dates: First submitted 2021-05-28; First posted 2021-06-21 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Industry standard stimulation (Active Comparator): Industry standard stimulation settings
  Interventions: Other: Stimulation parameters
- Experimental stimulation (Sham Comparator): Experimental stimulation settings
  Interventions: Other: Stimulation parameters

INTERVENTIONS:
Other: Stimulation parameters — Different device stimulation parameters

SUMMARY:
The objective of this study is to determine the efficacy of neuromodulation using various stimulation paradigms in the treatment of several disorders including chronic pain.

DETAILED DESCRIPTION:
Different stimulation parameters will be tried in a blinded fashion to compare efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for, and have been consented for, implantation of a neuromodulation device.

Exclusion Criteria:

* Non-English speaking

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in baseline pain measures | 6 months
  Pain outcomes measured using visual analogue scale

SECONDARY OUTCOMES:
Effect of stimulation on quality of life | 6 months
  As measured using EQ-5D-3L

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No